CLINICAL TRIAL: NCT00380796
Title: A Multicenter, Observational Study of the Long-term Safety of Infliximab (REMICADE) in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD). RESULTS COPD: REMICADE Safety Under Long Term Study in COPD
Brief Title: A Long-term Safety Study of Infliximab in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Type: Observational
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012292; C0168T70 (Other: Centocor)
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: COPD; Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: Collection of safety data for Cohort 1

INTERVENTIONS:
Drug: Collection of safety data for Cohort 1 — Twice-yearly collection of information about cancer incidence and cause of death among patients who participated in clinical trials of infliximab in the treatment of COPD. The follow-up period is 5 years.

SUMMARY:
The purpose of this long-term observational study is designed to collect additional information on incidence of cancer and cause of death among patients who have participated in clinical trials of infliximab in the treatment of COPD. Patients must have received at least 1 dose of study agent (ie, placebo or infliximab) in the primary studies to be eligible for participation in this long-term follow-up study. Information on deaths and cancers will be collected twice yearly for a period of 5 years from each patient's last safety visit in the primary study.

DETAILED DESCRIPTION:
This study is designed to collect long-term safety information on infliximab, from patients with COPD who participated in research studies using this drug. The primary COPD studies include C0168T54 (in the U.S.) and two small studies in Europe (EU0016 C0168X09 and EU0073 C0168X57). All patients who had at least one dose of study drug in those studies are being asked to participate in this long-term safety follow-up study which will provide important information about the study drug. The long-term effect of the study drug on new cancers and survival will be evaluated from data collected over a 5-year period which begins from each patient's last safety visit in the primary study. Data for this study will be collected at study entry and twice yearly thereafter up to a maximum of 5 years from each patient's last safety visit in the primary study. The last safety visit in the primary study is defined as the last visit for each subject during which adverse events (AEs)s are recorded in the primary study.Twice yearly, all participating study sites will be reminded to complete the electronic charts for each participating patient. At study entry, the following will be performed: (1) Medical history and physical examination, including ear, nose, and throat (ENT) examination performed by a qualified physician; (2) Chest x-ray(posterior and lateral), unless performed within 3 months prior to enrollment and (3) CT (computer imaging) scan of the chest (spiral preferred), unless performed within 6 months prior to enrollment. In addition, data will be collected at study entry on the use of commercial infliximab or any other anti-tumor necrosis factor (anti-TNF) agent subsequent to the last safety visit in the primary study. At each patient's subsequent visit, data will be collected by either direct contact with the patient (office visit or telephone call), review of patient's medical records, contact with the patient's primary care physician or oncologist. At the final visit (5 years from each patient's last safety visit in the primary study), the following will be performed: (1) Medical history and physical examination, including ENT examination performed by a qualified physician; (2) Chest x-ray, unless performed within the previous 3 months, and (3) CT scan of the chest (spiral preferred), unless performed within the previous 6 months.

The primary outcome of this study is Number of patients with each of the following safety events: malignancy or death. The secondary outcome of this study is the number of patients with malignancies by malignancy type (ie, Hodgkin's lymphoma, non-Hodgkin's lymphoma, head and neck cancers, lung cancer, other malignancies). No drug is provided

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been enrolled in previously completed clinical studies of infliximab in the treatment of COPD that are targeted for long term safety follow-up (ie, primary studies). Primary studies are defined as studies that have evaluated infliximab on an investigational basis and that have been identified by Centocor or health authorities as requiring long-term safety follow-up. These include Centocor protocol C0168T54, conducted in the USA, and 2 smaller studies conducted in the Netherlands (EU0016 C0168X09 and EU0073 C0168X57). Patients must have received at least one dose of study agent to be eligible.

Exclusion Criteria:

* Patients who are unwilling to respond to requests for long-term safety information will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who had at least one dose of study drug in clinical studies of infliximab in the treatment of COPD, that are targeted for long-term safety follow-up and were asked to participate in this long-term safety follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (26):
- United States (26):
  - Anaheim, California
  - San Diego, California
  - Bay Pines, Florida
  - Clearwater, Florida
  - Blue Ridge, Georgia
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Endwell, New York
  - Larchmont, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Easton, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greer, South Carolina
  - Spartanburg, South Carolina
  - Amarillo, Texas
  - Dallas, Texas
  - Salem, Virginia
  - Madison, Wisconsin